CLINICAL TRIAL: NCT00913042
Title: Assessment of New Blood Culture Methods on the Microbiological Documentation of Febrile Neutropenia
Acronym: HEMATOCPLUS
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: CRC 06021
Record Dates: First submitted 2009-06-02; First posted 2009-06-03 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2009-04

CONDITIONS: Febrile; Neutropenia; Post-chemotherapy
Keywords: Febrile neutropenia; Blood culture; Bacteremia; Bacterial DNA testing
MeSH Terms: conditions — Fever; Neutropenia; Febrile Neutropenia; Bacteremia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — bacterial inoculum in the blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: febrile neutropenia patient
  Interventions: Other: sample blood

INTERVENTIONS:
Other: sample blood — * Early culture
  * Bacterial DNA tests in blood

SUMMARY:
Febrile neutropenia are microbiologically documented in only 30% of the cases, and almost exclusively by blood cultures. The reasons for this low documentation are likely multiple: (1) some of these fevers are of non-infectious origin. (2) The bacterial inoculum present in the blood may be low and consequently undetectable by conventional blood cultures.

The primary objective of the study is to assess new blood culture procedures and technics, in order to improve the diagnostic yield of blood cultures during febrile neutropenic episodes.

DETAILED DESCRIPTION:
Evaluation criteria are 1) proportion of microbiologically documented infections 2) time elapsed from bed side sampling to microbiological diagnostic, in case of positive sample.

The assessed procedures included a large volume of blood, an early incubation made possible by the availability of a culture device in the hematology department, an early warning in case of positive blood culture, bacterial DNA detection in blood, and an early identification of the positive strains and their resistance profile.

We hypothesize that the combination of these different procedures will improve the proportion of microbiologically blood culture from 30 to 45%. One hundred and 20 episodes of febrile neutropenia are necessary to achieve this goal.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 y
* first episode of febrile neutropenia during a given neutropenic phase
* PMN < 500/mm3, chemotherapy-induced
* fever > 38°C twice, or < 38°3C once
* signed informed consent

Exclusion Criteria:

- patient already receiving empirical or therapeutic antibacterial after their first episode of febrile neutropenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Febrile neutropenia post-chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2008-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
proportion of microbiologically documented infections | Day 14 from inclusion

SECONDARY OUTCOMES:
clinical status at the end of hospitalisation | Day 30 from inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Pautas, PH, Principal Investigator — Henri Mondor University Hospital
Locations (1):
- Hematology Department, Paris 12 University Hospital Henri Mondor, Créteil, France